CLINICAL TRIAL: NCT06749912
Title: Effects of a Lower Back Wrap Device on Lower Back Pain, Physical Function, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Kyle Kelleran, Assistant Professor of Emergency Medicine, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008828
Record Dates: First submitted 2024-12-09; First posted 2024-12-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Lower Back Pain; Lower Back Pain Chronic; Acute Low Back Pain
Keywords: Low back pain; acute low back pain; symptom reduction; pain sensation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Lower back pain wrap (Experimental): During this arm the participants will wear the low back pain wrap device
  Interventions: Device: Low back pain wrap
- No device (No Intervention): No device will be used, but symptoms and function will be reported

INTERVENTIONS:
Device: Low back pain wrap — The low back pain wrap device includes heat, vibration, and red light to assist with reducing pain sensation, improving function.
  Arms: Lower back pain wrap

SUMMARY:
The goal of this counterbalanced cross-over study is to determine whether a recovery lumbar wrap effectively reduces lower back pain and improves outcomes related to physical function and quality of life in adults with LBP in adults 20-65 years old. This study will also explore whether improvements in other health metrics that are typically related to, or seen in, lower back pain research (i.e. stiffness, mobility, physical activity, validated clinical scoring methods, etc.) are improved with the use of the product.

The main question this study aims to answer is:

• Does the lumbar wrap effectively reduce low back pain symptoms and improve outcomes related to physical function and quality of life in adults with lower back pain.

Participants experiencing lower back pain will be asked to use the lower back wrap for at least 20-minutes per day for a 2-week period, counterbalanced with a 2-week period of no device use. Participants will fill out small daily surveys about their symptoms and complete a pre-, middle-, and post- survey and functional screening to determine efficacy of the device.

DETAILED DESCRIPTION:
Participants with both acute and chronic low back pain will be recruited from the emergency department, research registry, social media, and e-mails. Participants will be screened for inclusion and exclusion criteria and consented. This study utilizes a counterbalanced cross-over design. Each participant will complete both conditions: 1) Intervention (wrap), or 2) Control (Nothing). A counterbalanced assignment approach will be used to determine the starting condition for each participant (Phase 1). After completion of Phase 1, each participant will complete the remaining condition for Phase 2.

Each phase of the intervention will take 2 weeks, for a total of 4 weeks (2 weeks in Phase 1, 2 weeks in Phase 2). When participants are in the Intervention phase of the study, they will be asked to use the lower back wrap at least once per day for the standard treatment length (20 minutes). To support ecological validity, participants will be able to use the device ad libitum (several times throughout the day) as desired. The Researchers will administer simple daily surveys to log compliance to treatment.

A pre-, mid-, and post- survey and functional screening will be conducted to gather additional information about the participant and device efficacy and use.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 - 65
* Males and Females (50-50 split or close)
* Range of ethnicities
* Range of BMIs

Exclusion Criteria:

* Those with diagnosed cancer, infection, trauma, or LBP requiring surgical intervention
* Those currently undergoing rehabilitation treatment for LBP
* Those with other diagnosed conditions that may preclude them from safely participating
* Pregnant women
* Waist less than 26" or greater than 66" due to device limitations

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Pain | From enrollment to the end of treatment at 4 weeks
  Patients will report their level of pain daily and reflect on their pain over the past over the past 1-week at the start of the study and past 2-weeks during the follow-up surveys
  Pain Scale: 1-10, higher score = more pain.
Function survey | From enrollment to the end of treatment at 4 weeks
  Function will be assessed daily and every 2-weeks by survey.
Function test | From enrollment to the end of treatment at 4 weeks
  Function will be assessed every 2-weeks by a function screening via 5-repitition sit-to-stand.
  Function Scale: 5 point scale from "not at all" to "very much" indicating how much pain interfered with day-to-day activities.

SECONDARY OUTCOMES:
Medication usage | From enrollment to the end of treatment at 4 weeks
  Daily screening and every 2-weeks the participants will be asked about what prescription and over-the-counter medications, along with cannabis and THC, were used to help mediate the pain.
Other pain and rehabilitation use | From enrollment to the end of treatment at 4 weeks
  Participants will be surveyed daily and every 2-weeks about any other type of rehabilitation they used to help mediate their pain.
Device use- Frequency | For the 2-week device use period.
  Frequency of use will be recorded daily during the 2-week device intervention period
  Frequency scale: 0-5+ on a 6 point scale indicating how often the device was used per day.
Device use- Duration | For the 2-week device use period.
  Duration of use will be recorded daily during the 2-week device intervention period
  Scale: 2 point- default (20-minutes) or more. Free response in branching logic to insert amount of time if more than default.
Device use- Type | For the 2-week device use period.
  Type of use will be recorded daily during the 2-week device intervention period.
  Scale 1- How worn, gives options for under/over clothes & activity, resting, sitting, standing, ADLs, free response.

OTHER OUTCOMES:
Device use satisfaction | At the end of the 2-week device use period.
  At the conclusion of the 2-week device use period the participants will fill out a device satisfaction survey examining their experience with the device.
  25 question survey on how they felt the device worked. Most questions are on a 5-point Likert scale from "strongly agree" to "strongly disagree". The directionality changes based upon the question.
  Example:
  I could more easily complete daily tasks without pain during the study period when I used the device.
  1. Strongly Agree
  2. Agree
  3. Neither Agree nor Disagree
  4. Disagree
  5. Strongly Disagree

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Kelleran, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No